CLINICAL TRIAL: NCT02171910
Title: Doxapram as an Additive to Propofol Sedation in Sedation for Endoscopic Retrograde Cholangiopancreatography
Brief Title: Doxapram as an Additive to Propofol Sedation in Sedation for ERCP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jarno Jokelainen, MD, Senior physician, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Doxa1
Record Dates: First submitted 2014-06-15; First posted 2014-06-24 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Sedation; Hypoxia
Keywords: Cholangiopancreatography, Endoscopic Retrograde; Sedation
MeSH Terms: conditions — Hypoxia | interventions — Doxapram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doxapram (Active Comparator): Propofol sedation with a doxapram 1mg/kg i.v. bolus at induction and an i.v. infusion 1mg/kg/h) during the procedure
  Interventions: Drug: Doxapram
- Placebo (Placebo Comparator): Propofol sedation with a placebo i.v. bolus at induction and a placebo i.v. infusion during the procedure
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxapram
  Other Names: Dopram; Stimulex; Respiram
  Arms: Doxapram
Drug: Placebo — An injection and infusion of normal saline (NaCl 0.9%) as a placebo comparator to doxapram
  Arms: Placebo

SUMMARY:
Sedation is needed in order to complete endoscopic retrograde cholangiopancreatography (ERCP) to alleviate discomfort and pain during the procedure. This is usually achieved with use of opioids and/or sedative agents such as benzodiazepines or propofol. Traditionally benzodiazepines have been used but nowadays propofol is becoming the drug of choice for sedation during ERCP.

The problem with propofol sedation is the fact that it may case cardiorespiratory depression and there is no antidote for this like there is for benzodiazepines. Cardiovascular depression can usually be easily counteracted with drugs that are used to raise blood pressure or heart rate during general anesthesia but respiratory depression remains a problem.

The aim of this study is to try to counteract the respiratory depression caused by propofol sedation using an old respiratory stimulant doxapram as opposed to placebo using a double blind randomized protocol.

The investigators hypothesis is that boluses and an infusion of doxapram will alleviate the respiratory depression caused by propofol sedation.

ELIGIBILITY:
Inclusion Criteria:

* < 75 year of age
* Having ERCP
* Agrees to take part in the study

Exclusion Criteria:

* >75 years of age
* allergy to propofol or doxapram
* epilepsy
* Chronic Obstructive Pulmonary disease (COPD)
* Coronary artery disease (symptomatic)
* alcoholism
* declines to take part in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in arterial oxygenation | values recorded before the procedure, during the procedure at 5 min intervals and at the end of the procedure, on arrival at the recovery room and at 5 min, 10 min, and after that at 10 min intervals until discharge to ward
  Hypoxemia, oxygen saturation by pulse oximetry (SpO2 <90%), considered as a significant change

SECONDARY OUTCOMES:
change in systolic arterial pressure | values recorded before the procedure, during the procedure at 5 min intervals and at the end of the procedure, on arrival at the recovery room and at 5 min, 10 min, and after that at 10 min intervals until discharge to ward
  A drop of systolic arterial pressure to <90 mmHg is considered significant
Pulse (heartbeats/minute) | values recorded before the procedure, during the procedure at 5 min intervals and at the end of the procedure, on arrival at the recovery room and at 5 min, 10 min, and after that at 10 min intervals until discharge to ward
breathing rate (breaths/minute) | values recorded before the procedure, during the procedure at 5 min intervals and at the end of the procedure

OTHER OUTCOMES:
Sedation scales | values recorded before the procedure, during the procedure at 5 min intervals and at the end of the procedure
  Modified observer's assessment of Alertness/sedation (MOAA(S) and Bispectral Index (BiS)
End-tidal carbon dioxide (CO2) | values recorded before the procedure, during the procedure at 5 min intervals and at the end of the procedure
  A sampling catheter is placed in the nostril
Patient satisfaction | in the recovery room before discharge to ward
  The patient is asked to rate satisfaction to the given sedation on a seven step scale ranging from extremely dissatisfied to extremely satisfied
operating physician satisfaction | at the end of the procedure
  The operating physician is given a questionnaire and rates the following on a 4 step scale each: ease of applying the endoscope, patient co-operation, gagging/vomiting, coughing, belching, distracting movement of the patient. Also difficulty of the procedure is rated on a three step scale

CONTACTS AND LOCATIONS:
Overall Officials: Jarno Jokelainen, M.D., Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Uusimaa, Finland

REFERENCES:
- [Derived] Jokelainen J, Belozerskikh A, Mustonen H, Udd M, Kylanpaa L, Lindstrom O, Mazanikov M, Poyhia R. Doxapram as an additive to propofol sedation for endoscopic retrograde cholangiopancreatography: a placebo-controlled, randomized, double-blinded study. Surg Endosc. 2020 Dec;34(12):5477-5483. doi: 10.1007/s00464-019-07344-2. Epub 2020 Jan 28. PMID 31993819